CLINICAL TRIAL: NCT02442583
Title: Reducing Sedentary Behaviors Among Colorectal Cancer Survivors: Cancer Survivorship Center Pilot Project
Brief Title: Reducing Sedentary Behaviors Among Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00060174
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; survivor; exercise; physical activity; sedentary
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Phase 1, Step 1 (No Intervention): In this part, 15 early stage colorectal cancer survivors will fill out surveys and have a recorded phone interview regarding their physical activity and sedentary behaviors, to inform the creation of a brochure about sedentary behaviors.
- Arm 2: Phase 1, Step 2 (No Intervention): 5 early stage colorectal cancer survivors will have recorded telephone interviews to provide feedback about the brochure.
- Arm 3: Phase 2 (Experimental): 15 early stage colorectal cancer survivors will complete a baseline survey about sedentary behaviors, then wear an Actigraph device and self-report their sedentary activities for one week. They will receive feedback regarding their activity, and one month after receiving the feedback will participate in a phone survey regarding use of the brochure, physical activity and sedentary behaviors.
  Interventions: Other: Brochure regarding sedentary behavior

INTERVENTIONS:
Other: Brochure regarding sedentary behavior — This pilot will occur in two phases. Phase 1 will occur in two steps. In Step 1, we will conduct one-on-one telephone interviews with 15 early stage CRC (colorectal cancer) survivors to obtain their knowledge and insights about sedentary behaviors and ways to reduce them. Their input will be used to help create a brochure on sedentary behaviors. In Step 2, we will conduct one-on-one telephone interviews with 5 early stage CRC survivors to provide feedback about the brochure. In Phase 2, we will recruit 15 CRC survivors. After completing a baseline survey, they will be asked to both wear an ActiGraph and self-report their daily sedentary behaviors for one week. They will receive tailored feedback as to their average weakly levels of sedentary behaviors and receive the brochure. One month post-intervention, they will be asked to take part in telephone survey assessing sedentary behaviors, PA (physical activity), and use of brochure.
  Arms: Arm 3: Phase 2

SUMMARY:
Interview colorectal cancer survivors and use this input to create a brochure intended to guide reduction of sedentary behaviors in this population. Have colorectal cancer survivors review and comment on a draft of the brochure. A third group of colorectal cancer survivors will wear an Actigraph activity monitor for one week, then receive feedback on their activity level with the brochure. After one month this group will be surveyed by telephone regarding their use of the brochure, and their physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Early (stage 1 or 2) colorectal cancer
* 6 months or greater post treatment
* Does not follow guidelines for physical activity
* Average at least 6 hours a day of sedentary behaviors

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the print brochure, as measured by Likert scale. | Baseline
  Feasibility will be based in part on achieving higher (>5) on the Likert scale on topics such as usefulness, clarity, understanding how to use the materials.
Change in number of minutes per day of light to strenuous physical activity. | Baseline and 1 month
  The means and variances of self-reported total minutes per day of light to strenuous physical activity will be computed and compared from the survey at baseline, to the survey at the 1 month time point.
Change in number of minutes per day of bouts of sedentary behaviors. | Baseline and 1 month
  The means and variances of self-reported total minutes per day of sedentary behaviors, will be computed and compared from the survey at baseline, to the survey at the 1 month time point. Time per day will also be analyzed by type of activity.

SECONDARY OUTCOMES:
Covariation between baseline use of an ActiGraph, and self-reporting of sedentary behaviors | Baseline and 1 week
  To assess the baseline reliability of self-report, we will calculate the Pearson product-moment correlation coefficient between the self-report measure (total time and by each activity reported) and ActiGraph based on daily repeated measures for one week.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States